CLINICAL TRIAL: NCT03533101
Title: Tocilizumab for Cytokine Release Syndrome Prophylaxis in Peripheral Blood Haploidentical Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide
Brief Title: Tocilizumab for Cytokine Release Syndrome Prophylaxis in Haploidentical Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HE18-00010
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Cytokine Release Syndrome; Stem Cell Transplant Complications
Keywords: Tocilizumab; Haploidentical; Peripheral blood
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Adaptive design using two different doses of tocilizumab prophylaxis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab 4 mg/kg (Experimental): Tocilizumab 4 mg/kg IV single dose day -1 prior to haploidentical transplantation
  Interventions: Drug: Tocilizumab
- Tocilizumab 8 mg/kg (Active Comparator): Tocilizumab 8 mg/kg IV single dose day -1 prior to haploidentical transplantation
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — IL-6 receptor antibody pre-transplant administration to avoid cytokine release syndrome
  Other Names: Actemra; RoActemra

SUMMARY:
Tocilizumab will be administered prior to transplantation in order to prevent the onset of cytokine release syndrome and its complications associated to peripheral blood haploidentical hematopoietic stem cell transplantation with post-transplant cyclophosphamide

DETAILED DESCRIPTION:
Cytokine release syndrome (CRS) is a common and potentially severe toxicity associated to haploidentical peripheral blood (PBSC) hematopoietic stem cell transplantation (Haplo-HSCT), which was described previously in the context of immunotherapies for acute lymphoblastic leukemia such as chimeric antigen receptor T-cells and blinatumomab.

CRS is characterized by immune system activation with a high level of circulating inflammatory cytokines including IL-6. Haplo-HSCT recipients have a high incidence of post-transplant fever, with elevated IL-6 in absence of documented infection. CRS occurs more frequently when using PBSC, and severe cases have been associated to delayed engraftment, increased transplant-related mortality and lower survival.

Tocilizumab an IL-6 receptor-targeted monoclonal antibody has been effectively used to treat CRS in several scenarios, including Haplo-HSCT. Therefore, there is considerable interest for the development of a successful strategy for CRS prevention with tocilizumab, potentially eliminating complications. However, it is currently unknown whether the use of this monoclonal antibody can adversely affect the outcome of Haplo-HSCT recipients.

ELIGIBILITY:
Inclusion Criteria:

* Haploidentical transplant recipients
* Informed consent signature
* Previous diagnosis of any neoplastic, metabolic or autoimmune disease

Exclusion Criteria:

* History of immune deficiency virus infection
* Hepatitis C or B virus infection
* Documented bacterial of fungal infection prior to tocilizumab infusion
* Previous use of tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Cytokine release syndrome | 1 week
  Incidence of fever in the first seven days after haploidentical transplantation

SECONDARY OUTCOMES:
Hospitalization rate | 1 week
  Incidence of hospitalization in the first seven days after haploidentical transplantation
Adverse effects | 1 week
  According to Common Terminology Criteria for Adverse Events v5.0
IL-6 concentration | 1 week
  Concentration of serum IL-6 prior and during the first week after transplantation|

CONTACTS AND LOCATIONS:
Overall Officials: David Gómez-Almaguer, MD, Study Director — Hospital Universitario "Dr. José Eleuterio González"
Locations (1):
- Hospital Universitario Dr. Jose E Gonzalez UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka T, Narazaki M, Kishimoto T. Immunotherapeutic implications of IL-6 blockade for cytokine storm. Immunotherapy. 2016 Jul;8(8):959-70. doi: 10.2217/imt-2016-0020. PMID 27381687
- [Background] Teachey DT, Grupp SA. Cytokine Release Syndrome after Haploidentical Stem Cell Transplantation. Biol Blood Marrow Transplant. 2016 Oct;22(10):1736-1737. doi: 10.1016/j.bbmt.2016.08.010. Epub 2016 Aug 16. No abstract available. PMID 27543158
- [Background] Raj RV, Hamadani M, Szabo A, Pasquini MC, Shah NN, Drobyski WR, Shaw BE, Saber W, Rizzo JD, Jerkins J, Fenske TS, D'Souza A, Dhakal B, Zhang C, Konings S, Hari PN, Chhabra S. Peripheral Blood Grafts for T Cell-Replete Haploidentical Transplantation Increase the Incidence and Severity of Cytokine Release Syndrome. Biol Blood Marrow Transplant. 2018 Aug;24(8):1664-1670. doi: 10.1016/j.bbmt.2018.04.010. Epub 2018 Apr 19. PMID 29680516
- [Result] Abboud R, Keller J, Slade M, DiPersio JF, Westervelt P, Rettig MP, Meier S, Fehniger TA, Abboud CN, Uy GL, Vij R, Trinkaus KM, Schroeder MA, Romee R. Severe Cytokine-Release Syndrome after T Cell-Replete Peripheral Blood Haploidentical Donor Transplantation Is Associated with Poor Survival and Anti-IL-6 Therapy Is Safe and Well Tolerated. Biol Blood Marrow Transplant. 2016 Oct;22(10):1851-1860. doi: 10.1016/j.bbmt.2016.06.010. Epub 2016 Jun 16. PMID 27318038
- [Result] Kennedy GA, Varelias A, Vuckovic S, Le Texier L, Gartlan KH, Zhang P, Thomas G, Anderson L, Boyle G, Cloonan N, Leach J, Sturgeon E, Avery J, Olver SD, Lor M, Misra AK, Hutchins C, Morton AJ, Durrant ST, Subramoniapillai E, Butler JP, Curley CI, MacDonald KPA, Tey SK, Hill GR. Addition of interleukin-6 inhibition with tocilizumab to standard graft-versus-host disease prophylaxis after allogeneic stem-cell transplantation: a phase 1/2 trial. Lancet Oncol. 2014 Dec;15(13):1451-1459. doi: 10.1016/S1470-2045(14)71017-4. Epub 2014 Nov 14. PMID 25456364
- [Result] Drobyski WR, Szabo A, Zhu F, Keever-Taylor C, Hebert KM, Dunn R, Yim S, Johnson B, D'Souza A, Eapen M, Fenske TS, Hari P, Hamadani M, Horowitz MM, Rizzo JD, Saber W, Shah N, Shaw B, Pasquini M. Tocilizumab, tacrolimus and methotrexate for the prevention of acute graft-versus-host disease: low incidence of lower gastrointestinal tract disease. Haematologica. 2018 Apr;103(4):717-727. doi: 10.3324/haematol.2017.183434. Epub 2018 Jan 19. PMID 29351985